CLINICAL TRIAL: NCT03722888
Title: Development of a Videogame Prototype Targeting Cigarette and Marijuana Smoking, and Tobacco Product Prevention Among Young Adolescents
Brief Title: Development of a Videogame Prototype Targeting Cigarette and Marijuana Smoking, and Tobacco Product Prevention Among Young Adolescents (smokeScreen)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 140103293_IV
Record Dates: First submitted 2018-10-23; First posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Intervention Model Description: single group study with pre-post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adolescents who have previously smoked (Experimental): Adolescents given a pre-post survey to measure the effect of the game and building that into the smokeSCREEN video game to anonymously collect information on players' perspectives, beliefs, behaviors around smoking, and collaborating with youth programs to pilot test how the game can be implemented in real world settings.
  Interventions: Device: smokeSCREEN video game

INTERVENTIONS:
Device: smokeSCREEN video game — smokeSCREEN video game is web-based videogame intervention focused on tobacco use prevention in teens. The game has 1.5-2 hours of unique game play and focuses on combustible cigarettes, e-cigarettes, and flavored tobacco products.smokeSCREEN. Guided by the social cognitive theory and the theory of planned behavior, smokeSCREEN addresses a range of challenges that teens often face involving peer pressure and the use of tobacco products. Participants are provided access to the smokeSCREEN game through a private, password-protected website link and instructed to complete the game.

SUMMARY:
The goal of this sub-study is to learn more about how an educational videogame can feasibly be implemented and disseminated in youth programs.

DETAILED DESCRIPTION:
The specific aims of this sub-study are:

Specific Aim #1: Work with game development team to develop a web-based version of smokeSCREEN.

Specific Aim # 2: Build a pre-post survey into the smokeSCREEN game to anonymously collect survey information on players' perspectives, beliefs, behaviors around smoking.

Specific Aim # 3: Collaborate with youth programs to pilot test the implementation of the new web-based version of smokeSCREEN into youth programs.

ELIGIBILITY:
Inclusion Criteria:

* Include individuals who have smoked a cigarette previously (since we are evaluating the use of tobacco products in this study, we are including individuals who have previously smoked a cigarette)
* Willing to sit at a computer/tablet/smartphone and play a video game for 45-60 minutes and answer questions before and after playing the video game.
* Be enrolled in a youth program that we have a partnership with.

Exclusion Criteria:

* Does not fit the inclusion criteria.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
To determine the impact of a web-based prevention videogame intervention prototype, smokeSCREEN, on participants' beliefs involving tobacco product use - pre test survey. | baseline
  Participants completed a pre-survey through a secured, data collection website (Qualtrics Data Collection Software) and then played the videogame intervention. Fourteen questions were designed from the National Youth Tobacco Survey (2014)13 that focused on beliefs about cigarettes, e-cigarettes, and flavored tobacco were used. For beliefs, questions had 4-5 choices ranging from strongly disagree to strongly agree or definitely yes to definitely not, or 5 response choices ranging from very unlikely to very likely.
To determine the impact of a web-based prevention videogame intervention prototype, smokeSCREEN, on participants' beliefs involving tobacco product use - post test survey. | immediately after game play is completed
  Participants completed a post-survey through a secured, data collection website (Qualtrics Data Collection Software), after they have played the videogame intervention. Fourteen questions were designed from the National Youth Tobacco Survey (2014)13 that focused on beliefs about cigarettes, e-cigarettes, and flavored tobacco were used for the survey. For beliefs, questions had 4-5 choices ranging from strongly disagree to strongly agree or definitely yes to definitely not, or 5 response choices ranging from very unlikely to very likely.
To determine the impact of a web-based prevention videogame intervention prototype, smokeSCREEN, on participants' knowledge involving tobacco product use - pre test survey. | baseline
  Participants completed a pre-survey through a secured, data collection website (Qualtrics Data Collection Software), played the videogame intervention. Fourteen questions were designed from the National Youth Tobacco Survey (2014)13 that focused on knowledge about cigarettes, e-cigarettes, and flavored tobacco were used for the surveys. For knowledge, questions had 3 response choices (yes, not, and not sure).
To determine the impact of a web-based prevention videogame intervention prototype, smokeSCREEN, on participants' knowledge involving tobacco product use - post test survey. | immediately after game play is completed
  Participants completed a post-survey through a secured, data collection website (Qualtrics Data Collection Software), played the videogame intervention. Fourteen questions were designed from the National Youth Tobacco Survey (2014)13 that focused on knowledge about cigarettes, e-cigarettes, and flavored tobacco were used for the surveys. For knowledge, questions had 3 response choices (yes, not, and not sure).

SECONDARY OUTCOMES:
To collect data on participants' gameplay experience and satisfaction. | immediately after game play is completed
  The post-test survey included an additional 5 items on game experience and satisfaction from items designed for a previous videogame study on sexual risk reduction in young adolescents (e.g., "I would tell my friends to play this game," 4 response choices, ranging from strongly disagree to strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Fiellin, MD, Study Director — Yale University
Locations (3):
- United States (3):
  - Hamden Youth Center, Hamden, Connecticut
  - Leadership, Education, and Athletics Partnership (LEAP) Inc., New Haven, Connecticut
  - Farnam Neighborhood House, New Haven, Connecticut